CLINICAL TRIAL: NCT07219108
Title: The TAVERN Trial: Transcutaneous Auricular Vagus Enhanced Recovery in the NeuroICU - A Study of Clinical Outcomes and Cost Reduction
Brief Title: Transcutaneous Auricular Vagus Enhanced Recovery in the NeuroICU
Acronym: TAVERN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202507232
Record Dates: First submitted 2025-10-01; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute Neurological Injury; Acute Medical Conditions
Keywords: vagal nerve stimulation; pathologic process; acute medical condition; brain diseases; central nervous system diseases; spine cord injury; vascular diseases; hemorrhage; acute neurological condition
MeSH Terms: conditions — Pathologic Processes; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either stimulation or sham stimulation arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants will be fitted with an auricular stimulator, but blinded to whether they are receiving stimulation or not. Outcome scores and measures will be assessed and recorded by clinicians and research team members blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Auricular VNS Stimulation (Experimental): Participants receive twice-daily auricular vagal nerve stimulation
  Interventions: Device: Auricular Vagus Nerve Stimulation
- Sham Auricular VNS Stimulation (Sham Comparator): Participants will have an auricular vagal nerve stimulator placed in their ear twice daily, without the stimulation applied
  Interventions: Device: Sham Auricular Vagus nerve Stimulation

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation — Transcutaneous auricular vagal nerve stimulation
  Arms: Auricular VNS Stimulation
Device: Sham Auricular Vagus nerve Stimulation — Transcutaneous auricular vagal nerve ear clip applied without current/stimulation
  Arms: Sham Auricular VNS Stimulation

SUMMARY:
This study will demonstrate the impact of taVNS on reducing adverse events in NeuroICU patients, determine if taVNS reduces length of stay, and quantify the economic benefits of taVNS implementation in a broader neurocritical care population.

DETAILED DESCRIPTION:
Vagal nerve stimulation (VNS) has been studied as a novel method of reducing inflammation, and it has been successfully used in animal models of inflammatory conditions. The purpose of the proposed study is to determine if transcutaneous auricular VNS will impact 1) the occurrence of hospital-acquired infections, 2) the need for tracheostomy due to prolonged intubation, 3) the effect on hospital-stay physiology (e.g., vital signs and blood glucose metrics), and 4) inflammatory markers in the blood, and 5) the health economics.

This study will involve randomizing patients to stimulation with VNS, or sham stimulation. Blood samples for inflammatory marker analysis will be collected upon admission and serially throughout the patient's admission. Clinical events tracked during the hospital stay include the occurrence of hospital-acquired infections, tracheostomy, changes in vital signs and blood glucose, development of peri-hematomal edema, and interventions for edema (medical or surgical). Outcomes following admission will include intensive care unit and hospital stay, cost analysis of hospital stay, discharge destination, functional scores at discharge, and at follow-up visits for up to 1 year after discharge. No additional appointments will be made specially for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Admission to the NeuroICU within 36 hours of onset of an acute medical condition.
* Patient or authorized legal representative should be able to provide consent within 36 hours of ICU arrival
* Presence of at least one predictor of critical illness and/or severe brain / spinal cord injury:

  * Glasgow Coma Scale GCS >3 & <= 12 at admission
  * NIH stroke scale of 6 or greater
  * Requirement for ongoing mechanical ventilation
  * Requirement for ongoing vasopressor support
  * Diagnosis of subarachnoid hemorrhage
  * Diagnosis of intracerebral hemorrhage with hematoma volume > 5 ml
  * Diagnosis of moderate-severe traumatic brain injury (GCS >3 & <= 12)
  * Refractory Status epilepticus requiring continuous sedative infusions

Exclusion Criteria:

* Systemic immunosuppression
* Receiving ongoing cancer therapy
* Implanted electrical device (e.g., pacemaker, stimulator)
* Bradycardia on admission (Sustained bradycardia on arrival with a heart rate < 50 bpm for >5 minutes)
* Risk of imminent death or limitation of care (e.g., Glasgow Coma Scale of 3, pupillary dilatation)
* Expected ICU stay of less than 72 hours, as determined by attending physician or ICU fellow
* Pregnancy
* COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Assessment of the need for tracheostomy. | 14 days
  Quantification of patients who need tracheostomy due to prolonged intubation.
Occurrence of hospital-acquired infections | 14 days
  Data will be collected from medical records. Infections will include ventilator-associated pneumonia, catheter-associated urinary tract infections, bloodstream infection, clostridium difficile, and ventriculitis.
Changes in heart rate/heart trace | 14 days
  Evaluation of changes in centrally monitored heart rate/heart trace to calculate heart rate variability and QT interval.
Blood glucose measurement | 14 days
  Daily evaluation of blood glucose (mg/dL)
Insulin requirement | 14 days
  Assessment of daily insulin requirement (Units)
Hospital length of stay | Through hospital admission, average 14 days
  Total length of stay in the hospital, and in the intensive care unit
Neurological outcome | 1 year
  Modified Rankin Scale for Neurological Disability (minimum score 0, maximum score 6, better outcomes have lower scores)
Discharge destination | After hospital discharge, on average 14 days after admission.
  Patient discharge destination (ie, home, acute rehab)
Cost of ICU stay | Through hospital admission, average 14 days
  Evaluation of total ICU cost of stay ($)
Cost of Hospital Admission | Through hospital admission, average 14 days
  Evaluation of total hospital admission cost of stay ($)

SECONDARY OUTCOMES:
Change in the inflammatory markers TNF-α, IL-6, IL-10, and IFN-γ in plasma | 14 days
  Blood samples collected on days 1, 4, 7, 10, and 14 (Day 1 serves as baseline, prior to first treatment). Inflammatory markers will be reported in pg/mL.
Change in inflammatory markers in cerebrospinal fluid | 14 days
  rebrospinal fluid samples collected on days 1, 4, 7, 10, and 14 to evaluate for TNF-α, IL-6, IL-10, and IFN-γ . Inflammatory markers will be reported in pg/mL.
Cerebral Edema | 14 days
  Assessment of cerebral edema on each medically indicated and obtained head CT scan through assessment of selective sulcal volume (SSV)
Neurological outcome at discharge and first follow-up | up to 1 year.
  Disease-specific neurological outcome metric at discharge and first follow-up. Glasgow Coma Scale (GCS, maximum score: 15; minimum score: 3; better outcomes have higher scores).
Neurological Outcome at discharge and first follow-up | up to 1 year.
  Disease-specific neurological outcome metric at discharge and first follow-up. Glasgow Outcome Scale-Extended (GOSE, maximum score: 8; minimum score 1; better outcomes have higher scores).
Neurological Outcome at discharge and first follow-up | Up to 1 year.
  Disease-specific neurological outcome metric at discharge and first follow-up. Hemorrhagic stroke Glasgow Coma Scale (GCS, maximum score: 15; minimum score: 3; better outcomes have higher scores).
Neurological Outcome at discharge and first follow-up. | Up to 1 year.
  Disease-specific neurological outcome metric at discharge and first follow-up. National Institutes of Health Stroke Scale (NIHSS, maximum score: 42; minimum score: 1; better outcomes have lower scores).
Diagnosis of hospital-acquired infections | Through hospital admission, average 14 days
  Binary assessment of hospital-acquired infections (ventilator-associated pneumonia, catheter associated urinary tract infection, Clostridium difficile infection, ventriculitis) diagnosis acquired from hospital databases. (Yes or No rating, better outcomes associated with No).
Use of a ventilator | Through hospital admission, average 14 days
  Quantification of days on ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leuthardt, MD MBA, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan G, Huguenard AL, Donovan KM, Demarest P, Liu X, Li Z, Adamek M, Lavine K, Vellimana AK, Kummer TT, Osbun JW, Zipfel GJ, Brunner P, Leuthardt EC. The effect of transcutaneous auricular vagus nerve stimulation on cardiovascular function in subarachnoid hemorrhage patients: A randomized trial. Elife. 2025 Jan 9;13:RP100088. doi: 10.7554/eLife.100088. PMID 39786346
- [Background] Huguenard A, Tan G, Johnson G, Adamek M, Coxon A, Kummer T, Osbun J, Vellimana A, Limbrick D Jr, Zipfel G, Brunner P, Leuthardt E. Non-invasive Auricular Vagus nerve stimulation for Subarachnoid Hemorrhage (NAVSaH): Protocol for a prospective, triple-blinded, randomized controlled trial. PLoS One. 2024 Aug 23;19(8):e0301154. doi: 10.1371/journal.pone.0301154. eCollection 2024. PMID 39178291
- [Background] Huguenard AL, Tan G, Rivet DJ, Gao F, Johnson GW, Adamek M, Coxon AT, Kummer TT, Osbun JW, Vellimana AK, Limbrick DD, Zipfel GJ, Brunner P, Leuthardt EC. Auricular Vagus Nerve Stimulation Mitigates Inflammation and Vasospasm in Subarachnoid Hemorrhage: A Randomized Trial. medRxiv [Preprint]. 2024 May 1:2024.04.29.24306598. doi: 10.1101/2024.04.29.24306598. PMID 38746275